CLINICAL TRIAL: NCT02514395
Title: Translation & Linguistic Validation of Knee and Osteoarthritis Outcome Score (KOOS) Questionnaire in Marathi Language: Cross Section Survey
Brief Title: Translation & Linguistic Validation of Knee and Osteoarthritis Outcome Score (KOOS) Questionnaire in Marathi Language
Status: Completed | Type: Observational
Sponsor: TPCT's Terna College of Physiotherapy (Other)
Responsible Party: Principal Investigator, DR. SWATI MESHRAM, asso.prof., TPCT's Terna College of Physiotherapy
Other Study IDs: 2
Record Dates: First submitted 2015-07-06; First posted 2015-08-03 (Estimated); Last update posted 2023-11-27 (Actual); Status verified 2023-11

CONDITIONS: Health-Related Quality Of Life
Keywords: linguistic validation; KOOS; Marathi translation

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Other: disability index administration -self report form — Final T12 version of KOOS was given to the participants by an assistant who was not involved with any prior procedure. At the same time SF- 36 v2[32] generic health measure was also handed over. Filled forms were collected by the same assistant. Next day participants were given another blank copy of Marathi KOOS T12 versions. Hence each participant filled three forms.

SUMMARY:
Background:

KOOS is a self -administered instrument which assesses the patient's opinion about the Knee associated problems. For now it is available in English & various other languages & is a complete instrument in itself.

In India it has been translated in Hindi so far. However, each province in this country has a unique language. Maharashtra is the second largest state in India and Marathi is the regional language of the communication. Since KOOS is a self-report measure, its translation in this local language was thought to be necessary. This disease specific measure which is originally designed for English speaking region when employed to non-English population needed to be translated with unique method to achieve a normative equivalence and linguistic validation.

Methods: After taking permission from KOOS web manager T1, T2, T12, B1 & B2 versions were formatted according to the guidelines laid down by AAOS for cross cultural adaptation of health status measure. T12 version was sent for the field testing. Total 32 subjects who met the eligibility criteria were Included in this study.

Results:

Statistical analysis for reliability with test re-test method suggested Perfect correlation (r =1) between day 1 & 2. A range of 0.83-0.54 co-relation co-efficient (r) demonstrated the validity of KOOS and its subscales when compared against the 8 different domains of SF-36. All this correlations were statistically highly significant. Sport and recreation subscale had many missing responses since many items in this subscale were not appropriate for the Maharashtrian cultural set-up. Participants additionally provided the information about other functional activities which were difficult to execute due to knee associated pain and disability.

Conclusion: Marathi version of KOOS is proved to be a reliable & valid measure. Future scope: this study demonstrate a need to undertake the cross cultural adaptation since a constant pattern of impairment revealed in the execution of daily activities such as sitting on the floor and attending certain yoga postures etc.

Key words: linguistic validation, disease specific self-report, KOOS, Marathi translation, quality of life.

DETAILED DESCRIPTION:
Disability index is used as the Outcome measures and is a diagnostic tools and prognostic tool. This index allows a healthcare professional to measure impact of psycho-social and physical factors on the functional performance, ability of the patient. The people suffering from osteoarthritis is determined by the interplay of psychosocial, physical and physiological neuromuscular factors such as Quadriceps strength, knee pain, and age . These components have shown to be more important determinants of functional impairment in elderly subjects than the severity of knee osteoarthritis as assessed radiographically.Disability index which are designed to measure the influence of this factors on functional outcome are hence used clinically to justify the treatment and capture the meaningful recovery.

The disease specific measures which are designed to assess the specific diagnostic group or specific population with a goal to detect a clinical change with the intervention of known efficacy should have good reliability, validity, responsiveness, and low burden of administration to be clinically useful. Such measures should be standardized and patient- centered that can be administered at a low cost. Hence a questionnaire was developed to assess short- and long-term patient-relevant outcomes following knee injury in form of Knee Injury and Osteoarthritis Outcome Score (KOOS). This is self-administered and assesses five outcomes: Pain, Symptoms, Activities of Daily Living, Sport and Recreation Function, and Knee-Related Quality Of Life.

The KOOS meets basic criteria of outcome measures and can be used to evaluate the course of knee injury and treatment outcome. KOOS has been used as a reliable and valid measure when used to evaluate the effectiveness of an intervention in knee osteoarthritis, total knee replacement anterior cruciate ligament and cartilage injury. It has been converted in various regional languages. KOOS has been translated in national language of India ie. Hindi. However, in many provinces of India the primary language of communication varies. In this multi-linguistic country the language shift happens in every province concordant with diversified culture. Maharashtra is second largest state in India with estimated population is over 117 million appx. the primary language of communication is Marathi and over 70 % of population communicate in this regional language. A need for the translational and cross cultural adaptation has been emphasized for the effective and reasonable measurement of responses to any self-report measure whenever and wherever applicable. This is true especially if the self-report measure which was originally designed for English speaking region is being employed to non-English population. It is difficult to achieve normative equivalence which is dependent on openness with strangers, political opinions, tendency to conform or assert oneself , since cultures differ on how willing they are to share personal information. On the other hand information relevant to semantic and conceptual equivalence of demographic questions across languages, can be extracted with less difficulty since the words and ideas are more general and commonly used. This emphasizes a need to translate a health status self-administered measure for use in a new country. It is now recognized that a unique method should be used to achieve a linguistic validation to reach equivalence between the original source and target language of the measure or instrument. A published report by ISPOR suggests the consensus on following Principles of Good Practice in translation and cultural adaptation of any self-report questionnaire. A guidelines has been evolved for the adaptation process and is available in form of a template. Adaptation process is designed to attain semantic, idiomatic, experiential, and conceptual equivalence between the source and target questionnaires Since KOOS is the self-administered instrument, its translation in this local language was thought to be necessary as the majority of population attending physiotherapy clinics communicates in Marathi. Unavailability of the Marathi versions of KOOS hence, poses a difficulty in functional evaluation in this population on day to day basis before and after the treatment. Hence, there exists a need to provide valid and reliable Marathi version of KOOS, so as to facilitate the better understanding of functional evaluation findings in population suffering from knee osteoarthritis. This study aims to translate and check the psychometric properties of the translated version of the KOOS as per the guidelines laid down by AAOS. Objective of this study is to provide a valid and reliable instrument in the regional language which intends to evaluate disease specific functional problems in Marathi speaking population.

Methods:

Study design: cross section survey design- a validation study. Permission was obtained from Institutional local ethic committee. This study was carried out in 2 phases.

Phase I consisted of translation of the English version of KOOS into the Marathi version. Second phase consisted of the field testing of the translated version to check test-retest reliability and validity.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects who were diagnosed for osteoarthritis of knee
2. who have not undergone any physical therapy treatment previously were considered eligible.

Exclusion Criteria:

1)subjects who didn't give any informed consent

Ages: 40 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Eligible subjects who the fulfilled the inclusion criteria were register for the study.
Sampling Method: Probability Sample
Enrollment: 32 (Actual)
Dates: Start 2012-09; Primary Completion 2013-07 (Actual); Study Completion 2013-11 (Actual)

PRIMARY OUTCOMES:
Knee Injury and Osteoarthritis Outcome Score (KOOS) | 2 days
  It is a questionnaire designed to assess short and long-term patient-relevant outcomes following knee osteoarthritis or mechanical knee somatic dysfunction.